CLINICAL TRIAL: NCT02992600
Title: Postoperative Cognitive Dysfunction: Correlations With Olfactory Dysfunction and Related Gene Changes
Status: Completed | Type: Observational
Sponsor: Han Yuan (Other)
Responsible Party: Sponsor-Investigator, Han Yuan, Physician in Anesthesiology, Xuzhou Medical University
Organization: Xuzhou Medical University (Other)
Other Study IDs: XYFY2016-KL018-01
Record Dates: First submitted 2016-12-02; First posted 2016-12-14 (Estimated); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: non-cardiac surgery; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples With DNA — blood

GROUPS / COHORTS (2):
- study group: 300 male and female patients undergoing non-cardiac surgery are enrolled at the Affiliated Hospital of Xuzhou Medical University [Jiangsu China]. Patients will be divided into POCD and non-POCD groups according to the scores of neuropsychological tests.
- control group: 30 healthy volunteers are enrolled for calculating the Z-scores of study group.

SUMMARY:
To study on the Postoperative Cognitive Dysfunction: Correlations With Olfactory Dysfunction and Related Gene Changes.To explore whether the olfactory dysfunction could be used as a predictor of POCD and to provide reference for POCD prevention, early detection and timely diagnosis and treatment.

ELIGIBILITY:
Inclusion criteria:

* Between 60 to 85 years old;
* Undergoing non-cardiac and non-neurological surgery under general anesthesia;
* Expected hospital stay ≥5 days;
* American Society of Anesthesiologists class I or II.

Exclusion criteria:

* Mental or neurodegenerative diseases;
* History of severe trauma or surgery within one year;
* History of nasal or sinus illness or surgery;
* Cold or influenza within 3 weeks;
* Significant history of organ dysfunction;
* Previous neuropsychological testing;
* Difficulty to perform tests (including severe visual or auditory disorders);
* Mini-Mental State Examination (MMSE) <24 points, <20 points if the participant only attended elementary school, or <17 points if the participant did not go to school.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We included 300 male and female patients undergoing non-cardiac surgery at the Affiliated Hospital of Xuzhou Medical University and 30 healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
the neuropsychological test battery to measure cognitive function | 1 day before surgery(baseline)
olfaction test to measure the sense of smell | 1 day before surgery(baseline)
the neuropsychological tests to measure cognitive function | within 5 to 10 days (average of 7 days) after surgery
olfaction test to measure the sense of smell | within 5 to 10 days (average of 7 days) after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia of the Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
within six months after the trial complete